CLINICAL TRIAL: NCT01619384
Title: Pyrosequencing to Identify Alterations in Intestinal Microbiota Following a Stress Reduction Course
Brief Title: Mindfulness-Based Stress Reduction and the Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRB# 00044
Record Dates: First submitted 2012-06-11; First posted 2012-06-14 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Posttraumatic Stress Disorder; Irritable Bowel Syndrome
Keywords: posttraumatic stress; irritable bowel
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Irritable Bowel Syndrome | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (No Intervention): Usual VA care
- MBSR (Experimental): participation in an 8-week stress reduction course (mindfulness-based stress reduction)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — An 8-week validated stress reduction program, designed to teach mindfulness.
  Arms: MBSR

SUMMARY:
This proposed study aims to determine whether decreasing stress levels in persons with posttraumatic stress disorder (PTSD) can lead to a change in the intestinal microbiota, assessed 8 weeks after enrollment.

DETAILED DESCRIPTION:
The gut microbiota is known to be integral to gastrointestinal health and disease. Psychological stress has been shown to significantly alter the gastrointestinal microbiota of rats, rhesus monkeys, and humans. These studies have consistently shown decreases in lactobacilli among other changes in species that correlate with an increase in diarrheal symptoms. While it is unclear whether stress causes diarrhea leading indirectly to a disruption in the native microbiota, or whether stress leads directly to changes in the microbiota that then lead to diarrhea; there is a growing body of evidence to support the latter. Differences in microbiota have also been shown to be present in irritable bowel syndrome (IBS) and predispose or protect against other forms of diarrhea including bacterial gastroenteritis and radiation-induced diarrhea. In addition, treatment with probiotics containing lactobacillus and other species has been shown to help alleviate IBS symptoms. Stress is hypothesized to act on the microbiota via the brain-gut axis through endocrine, immunological, and/or neurological pathways. This proposed study aims to determine whether decreasing stress levels in persons with posttraumatic stress disorder (PTSD) & IBS can lead to a change in the intestinal microbiota, assessed 3 weeks after enrollment. It also seeks to determine if a change in intestinal microbiota correlates with a decrease in IBS symptoms. We propose to use broad-range bacterial 16S rRNA gene PCR with 454 pyrosequencing to characterize the fecal microbiota and correlate changes in bacterial communities to IBS symptoms at baseline and after completion of an 8-week-stress reduction course in 15 patients with PTSD & IBS and to compare these findings to 5 patients with PTSD & IBS undergoing usual care without a stress-reduction course.

ELIGIBILITY:
Inclusion Criteria:

* posttraumatic stress disorder

Exclusion Criteria:

* psychosis
* suicidal ideation with intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in intestinal microbiome | baseline, 8 weeks, 4-month follow-up
  characterization of the intestinal microbiome is a primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: David Kearney, MD, Principal Investigator — Seattle Institute for Biomedical and Clinical Research
Locations (1):
- VA Puget Sound, Seattle, Washington, United States